CLINICAL TRIAL: NCT06145997
Title: Collecting Pragmatic Data Via Electronic Health Records: ACUAWARE Feasibility and Acceptability Study
Brief Title: Feasibility and Acceptability Study of ACUAWARE
Acronym: ACUAWARE
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: University of Utah (Other)
Collaborators: Pace University (Other)
Responsible Party: Sponsor
Other Study IDs: 00139124
Record Dates: First submitted 2023-11-12; First posted 2023-11-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Feasibility study; Acceptability study
MeSH Terms: conditions — Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with chronic pain: Standard acupuncture care will be provided to persons (n=50) with chronic pain. Standard care is defined as the care a participant was already receiving and that care will not be interrupted in any way for any study participant.
  Interventions: Other: Acupuncture therapy

INTERVENTIONS:
Other: Acupuncture therapy — Acupuncture therapy (AT) is delivered by Licensed Acupuncturists (LAcs). Treatment plans are determined according to each patient's presentation and resulting traditional East Asian medicine (TEAM) differential diagnosis. TEAM therapeutics include AT, Chinese herbal medicine (CHM), Kampo herbal medicine, gua sha, tui na, cupping and lifestyle advice. All TEAM therapeutics are allowed in this study because it is a pragmatic, effectiveness study.

SUMMARY:
This study aims to gather preliminary feasibility and acceptability data to justify a subsequent trial that would fill a gap in knowledge regarding acupuncture therapy (AT) effects on interoceptive awareness (IA) among those with chronic pain.

DETAILED DESCRIPTION:
This study aims to gather preliminary feasibility and acceptability data to justify a subsequent trial that would fill a gap in knowledge regarding acupuncture's effects on interoceptive awareness among individuals with chronic pain. Our primary hypotheses are that (1) Feasibility: it is feasible for us to enroll and retain 70% of the patients and it is feasible to collect data from at least 70% of participants at 3-months follow-up, and (2) Acceptability: it is acceptable for 70% of licensed acupuncturists to use Acu-Track Registry; it is acceptable for 70% of patients to complete questionnaires emailed to them via Acu-Track Registry.

The investigators propose to evaluate these hypotheses by conducting a prospective, pragmatic single-arm feasibility and acceptability study among individuals with chronic pain of any etiology or location, except if due to cancer. Chronic pain is defined as pain that persists or recurs for more than 3 months.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Age 18 or older;
* experiencing chronic pain,
* complaint of 3+ months,
* score of 5 or greater on a 1-10 scale;
* able to provide informed consent
* willing to sign an approved consent form that conforms to federal and institutional guidelines,
* English speaking and writing.

Exclusion Criteria:

Prior or current diagnosis of:

* cancer,
* Multiple Sclerosis (MS),
* any Dementia,
* Parkinson's Disease,
* Autism Spectrum Disorder,
* Pregnancy,
* Fibromyalgia,
* Eating Disorder,
* Down's Syndrome
* Schizophrenia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults in the United States with chronic pain, defined as pain lasting of 3 or more months, and given a score of 5 or greater on a 1-10 scale.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Feasibility metrics - rate of enrollment | 24 months
  Rate of enrollment of acupuncturists and patients (frequency count)
Feasibility metrics - rate of retention | 24 months
  Rate of retention of acupuncturists and participants (frequency count)
Feasibility metrics - rate of questionnaire completion | 24 months
  Rate of questionnaire completion by participants (frequency count)
Feasibility metrics - completion rate of acupuncture therapy | 24 months
  Rate of completion of acupuncture therapy (AT) (frequency count)
Feasibility metrics - rate of serious adverse events | 24 months
  Rate of serious adverse events (frequency count)
Acceptability metrics | 24 months
  Acceptability ratings by licensed acupuncturists and by participants. Acceptability is asked in a binary question: "Is it acceptable to you to use the Acu-Track registry?" Yes/No. We define "acceptable" as 70% or more of licensed acupuncturists to use Acu-Track Registry; and acceptable for 70% or more of patients to complete questionnaires emailed to them via Acu-Track Registry.

SECONDARY OUTCOMES:
Multidimensional Assessment of Interoceptive Awareness Scale, 2 (MAIA-2) | 24 months
  The MAIA-2, or Multidimensional Assessment of Interoceptive Awareness Scale, will be used to measure interoceptive awareness (IA). The MAIA-2 is comprised of 8 subscales and 37 items. Items are scored 0-5, with higher scores indicating increased IA.
Global Impression of Change (GIC) | 24 months
  This simple 1 question measure is a retrospective rating scale that asks the patient how much better or worse their health complaint is since beginning their course of treatments or care. It is a quick and straightforward way to gauge a patient's own belief about their improvement so far. Our PGIC scale is health complaint specific, rather than general, providing the ability to focus on monitoring a specific problem.
Physical Function from Patient-Reported Outcomes Measurement Information System Global-10 (PROMIS-10) | 24 months
  PROMIS-10 scoring will be used to evaluate physical function. PROMIS-10 scoring allows each of the individual items to be examined separately to provide specific information about perceptions of health (e.g., physical function, pain, fatigue, emotional distress, social health and general perceptions of health). We are using the single item: "To what extent are you able to carry out your everyday physical activities such as walking, climbing stairs, carrying groceries, or moving a chair?" Likert type scale 5-1: (5) completely, to (1) not at all.
Global Mental Health | 24 months
  PROMIS-10 scoring will also be used to evaluate global mental health. We are using the single item: "In the past 7 days: How often have you been bothered by emotional problems such as feeling anxious, depressed, or irritable?" Likert type scale 0-10: (0) no pain to (10) worst pain imaginable
Anxiety | 24 months
  PROMIS-10 scoring allows each of the individual items to be examined separately to provide specific information about perceptions of health. We are using the single item: "In the past 7 days: How often have you been bothered by emotional problems such as feeling anxious?" Likert type scale 0-10: (0) no pain to (10) worst pain imaginable.
Depression | 24 months
  PROMIS-10 scoring allows each of the individual items to be examined separately to provide specific information about perceptions of health. We are using the single item: "In the past 7 days: How often have you been bothered by emotional problems such as feeling depressed?" Likert type scale 0-10: (0) no pain to (10) worst pain imaginable.
Irritability | 24 months
  PROMIS-10 scoring allows each of the individual items to be examined separately to provide specific information about perceptions of health. We are using the single item: "In the past 7 days: How often have you been bothered by emotional problems such as feeling irritable?" Likert type scale 0-10: (0) no pain to (10) worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Taylor-Swanson, PHD, Principal Investigator — University of Utah College of Nursing
Locations (1):
- University of Utah College of Nursing, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be used or received in this study, thus no IPD can be made available to other researchers.

REFERENCES:
- [Background] Chou R, Deyo R, Friedly J, Skelly A, Hashimoto R, Weimer M, Fu R, Dana T, Kraegel P, Griffin J, Grusing S, Brodt ED. Nonpharmacologic Therapies for Low Back Pain: A Systematic Review for an American College of Physicians Clinical Practice Guideline. Ann Intern Med. 2017 Apr 4;166(7):493-505. doi: 10.7326/M16-2459. Epub 2017 Feb 14. PMID 28192793
- [Background] Di Lernia D, Serino S, Riva G. Pain in the body. Altered interoception in chronic pain conditions: A systematic review. Neurosci Biobehav Rev. 2016 Dec;71:328-341. doi: 10.1016/j.neubiorev.2016.09.015. Epub 2016 Sep 18. PMID 27654341
- [Background] Grissa MH, Baccouche H, Boubaker H, Beltaief K, Bzeouich N, Fredj N, Msolli MA, Boukef R, Bouida W, Nouira S. Acupuncture vs intravenous morphine in the management of acute pain in the ED. Am J Emerg Med. 2016 Nov;34(11):2112-2116. doi: 10.1016/j.ajem.2016.07.028. Epub 2016 Jul 20. PMID 27475042
- [Background] Teng B, Wang D, Su C, Zhou H, Wang T, Mehling WE, Hu Y. The multidimensional assessment of interoceptive awareness, version 2: Translation and psychometric properties of the Chinese version. Front Psychiatry. 2022 Nov 11;13:970982. doi: 10.3389/fpsyt.2022.970982. eCollection 2022. PMID 36440402